CLINICAL TRIAL: NCT02262182
Title: Evaluation of the Interest of Positive Expiratory Pressure (PEP) Delivery by EzPAP® Device Associated With Respiratory Physiotherapy in the Treatment of Postoperative Pulmonary Atelectasis in Patients After Cardiac Surgery
Brief Title: Interest of Positive Expiratory Pressure (PEP) Delivery by EzPAP® After Cardiac Surgery in the Management of Postoperative Atelectasis
Acronym: PEPKIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RC14_0033
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Pulmonary Atelectasis
Keywords: Atelectasis, Respiratory physiotherapy, end expiratory pressure, EzPAP®, cardiac surgery
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KP group (Experimental): PEP delivery by EzPAP® device with manual chest physiotherapy .
  Interventions: Other: KP group
- KM group (Placebo Comparator): Manual chest physiotherapy only;
  Interventions: Other: KM group

INTERVENTIONS:
Other: KP group
  Other Names: Associated to manual chest physiotherapy, patients receive twice a day 4 periods of PEP delivery by EzPAP® device during 25 respiratory cycles.
  Arms: KP group
Other: KM group
  Other Names: Patients of the control group benefit only from manual chest physiotherapy twice a day
  Arms: KM group

SUMMARY:
Pulmonary atelectasis is a frequent respiratory postoperative complication in cardiac surgery. Classically, the treatment of these patients is based on manual chest physiotherapy. Our objective is to evaluate the interest of association of positive end expiratory delivery sessions with the EzPAP® device. We perform a prospective monocentric, open label trial. Patients with atelectasis after scheduled cardiac surgery with cardiopulmonary bypass are included. They benefit from manual chest therapy and are randomised to receive or not positive end expiratory pressure sessions twice a day. The primary endpoint is the effect of this treatment on atelectasis radiological score after 2 days of treatment. The secondary endpoints are: oxygen saturation(SpO2)/inspired oxygen(FiO2) ratio, qualitative evaluation of ventilatory function, respiratory & cardiac rate, pain, inspiratory pressure (sniff test), patient satisfaction, duration of intensive care unit (ICU) and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in ICU after cardiac surgery by sternotomy with cardiopulmonary bypass presenting a pulmonary atelectasis after extubation, diagnosed by chest X-ray in postoperative period (day1 to day 2).
* Patients over 18 years of age
* Informed patient

Exclusion Criteria:

* Cardiac arrhythmia
* Hemodynamic instability (mean blood pressure < 65 mmHg or > 95 mmHg)
* Respiratory rate > 35/min
* Undrained pneumothorax
* Predictable trachea intubation or emergent surgery
* Patient oral refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Radiological atelectasis score | Day 2 post-inclusion
  This score was first described by Pasquina P et al in 2004

SECONDARY OUTCOMES:
Radiological atelectasis score | Days 1 and 3 post-inclusion
  This score was first described by Pasquina P et al in 2004
SpO2/FiO2 ratio | Days 1, 2 and 3 post inclusion
  This ratio is measured before and after session
Cardiac and respiratory rate | Days 1, 2 and 3 post inclusion
  Measurement performed at the same time as SPO2 (patients are monitored)
Qualitative evaluation of ventilatory function (nasal flaring, superficial tachypnea, use of accessory muscle, paradoxical abdominal respiration, cough difficulty) before and after session | Days 1, 2 and 3 post inclusion
  This respiratory function assessment is performed in a qualitative way
Dyspnea evaluation | Days 1, 2 and 3 post inclusion
  Dyspnea is measured with a visual analogue scale before and after session
Pain evaluation | Days 1, 2 and 3 post inclusion
  Pain is measured with a visual analogue scale before and after session
Vesicular murmur intensity | Days 1, 2 and 3 post inclusion
  Vesicular murmur absent = 0, reduce = 1, present and normal = 2 Intensity is measured with an electronic stethoscope before and after session
Inspiratory pressure measurement | Days 2 and 3 post inclusion
  This measurement (so called sniff test) is assessed with MicroRPM device before and after session
Assessment of patient satisfaction and tolerance of EzPAP device | Day 3 post inclusion
  A questionnaire of 10 answer with semi-quantitative scale

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes Universitary Hospital, Saint-Herblain, France